CLINICAL TRIAL: NCT04353271
Title: A Randomized Phase 2/3 Trial of Hydroxychloroquine In Covid-19 Kinetics
Brief Title: Trial of Hydroxychloroquine In Covid-19 Kinetics
Acronym: THICK
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: FDA recommendations to not use outside of the hospital setting or in a clinical trial due to the risk of cardiac arrhythmias
Sponsor: University of South Alabama (Other)
Responsible Party: Principal Investigator, William Richards, Professor and Chair Surgery, University of South Alabama
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: [1582736-1]
Record Dates: First submitted 2020-03-25; First posted 2020-04-20 (Actual); Results first posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Covid 19; Corona Virus Infection
Keywords: covid 19; plaquenil; hydroxychloroquine
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Randomized placebo verses medication clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded to subject and investigators
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hydroxychloroquine (Experimental): Subjects in this arm will receive the study drug
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator): Subjects in this arm will take placebo for 6 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine 800 mg initial dose then 6-8 hours later HCQ 600 mg, then 200 mg three times per day for 4 days.
  Other Names: plaquenil
  Arms: Hydroxychloroquine
Other: Placebo — Placebo take 4 tabs, then 6-8 hours later take 3 tabs, then take 1 tab three times per day for 4 days.
  Arms: Placebo

SUMMARY:
To test if the medication Hydroxychloroquine will decrease the amount of virus(as measured by PCR) , 7 days after initiation of therapy compared to control patients receiving placebo.

The study design is a randomized (5 days of medication v. 5 days of placebo) clinical trial initiated immediately after diagnosis in ambulatory health care workers at University of South Alabama Health, or in ambulatory USA patients. At 7 days after enrollment another nasopharyngeal swab will be taken to measure if the virus is still present. At 10 weeks we will measure immunity from Covid-19 using a single blood sample. It is a phase 2/3 clinical trial.

DETAILED DESCRIPTION:
Hydroxychloroquine (HCQ), which is a less toxic derivative of chloroquine (CQ), has been shown to be effective in inhibiting Covid-19 infection in vitro. The evidence from clinical research trials is sparse and has many flaws. Much of the Chinese experience with Chloroquine comes from a letter to the editor and a news briefing/conference held on February 15, 2020. The letter describes experience with more than 100 patients treated with CQ in multicenter clinical trials but the letter provides no quantitative data to back their claims. At least one non-randomized clinical trial has been performed in Europe. Covid-19 infected patients received 10 days of HCQ daily and underwent daily testing of viral loads from nasopharyngeal swabs. The subjects receiving HCQ were much more likely (P<0.02) to clear their viral load than subjects who did not receive HCQ. The study had many flaws, which make the conclusions less valuable than rigorously designed randomized clinical trial. This study is designed as a randomized, blinded trial to either confirm or refute the efficacy of HCQ in early treatment of Covid19 infection to ameliorate disease severity, and reduce viral load.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms occurring within 3 days prior to patient presenting to USA Facility for PCR nasopharyngeal swab
* Nasopharyngeal swab positive for Covid-19 infection and/or exposure and/or symptoms congruent with fever and cough
* Male or Female age 19 to 89 years
* Able to take oral medications
* Patients not requiring hospitalization
* Provision of informed consent

Exclusion Criteria:

* Known history of EKG QTc prolongation abnormality
* Contraindication or allergy to hydroxychloroquine
* Retinal eye disease
* Known glucose-6 phosphate dehydrogenase (G-6-PD) deficiency
* Known chronic kidney disease, stage 4 or 5 or receiving dialysis
* Weight < 40 kg
* Current use of: hydroxychloroquine or cardiac medicines of: flecainide, Tambocor; amiodarone, Cordarone, Pacerone; digoxin or Digox, Digitek, Lanoxin; procainamide or Procan, Procanbid, propafenone, Rythmal)
* Known hepatic disease (cirrhosis, hepatitis)
* Active treatment for cancer (chemotherapy, radiation, surgery within 3 months
* On immunosuppressive drugs steroids, antirejection medications.
* Recipient of solid organ transplant
* Pregnancy/breastfeeding
* Past medical history Porphyria (may exacerbate disease)
* PMH Psoariasis (can worsen disease)
* No access to internet or email
* Current suicidal thoughts according to Columbia scale
* In the screening process before signing consent, subjects will be asked if they are suicidal. If this response is yes, patients will be excluded from trial and directed to the National Suicide Prevention Lifeline: 1-800-273-8255.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William O Richards, MD, Principal Investigator — University of South Alabama College of Medicine
Locations (1):
- University of South Alabama, Mobile, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Percival I. Nuclear winter. Practitioner. 1988 Feb 8;232(1442):140-1. No abstract available. PMID 3217330
- [Background] Gao J, Tian Z, Yang X. Breakthrough: Chloroquine phosphate has shown apparent efficacy in treatment of COVID-19 associated pneumonia in clinical studies. Biosci Trends. 2020 Mar 16;14(1):72-73. doi: 10.5582/bst.2020.01047. Epub 2020 Feb 19. PMID 32074550
- [Background] Liu J, Cao R, Xu M, Wang X, Zhang H, Hu H, Li Y, Hu Z, Zhong W, Wang M. Hydroxychloroquine, a less toxic derivative of chloroquine, is effective in inhibiting SARS-CoV-2 infection in vitro. Cell Discov. 2020 Mar 18;6:16. doi: 10.1038/s41421-020-0156-0. eCollection 2020. No abstract available. PMID 32194981
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Background] Yao X, Ye F, Zhang M, Cui C, Huang B, Niu P, Liu X, Zhao L, Dong E, Song C, Zhan S, Lu R, Li H, Tan W, Liu D. In Vitro Antiviral Activity and Projection of Optimized Dosing Design of Hydroxychloroquine for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Clin Infect Dis. 2020 Jul 28;71(15):732-739. doi: 10.1093/cid/ciaa237. PMID 32150618
- [Background] Sahraei Z, Shabani M, Shokouhi S, Saffaei A. Aminoquinolines against coronavirus disease 2019 (COVID-19): chloroquine or hydroxychloroquine. Int J Antimicrob Agents. 2020 Apr;55(4):105945. doi: 10.1016/j.ijantimicag.2020.105945. Epub 2020 Mar 17. No abstract available. PMID 32194152
- [Background] Colson P, Rolain JM, Lagier JC, Brouqui P, Raoult D. Chloroquine and hydroxychloroquine as available weapons to fight COVID-19. Int J Antimicrob Agents. 2020 Apr;55(4):105932. doi: 10.1016/j.ijantimicag.2020.105932. Epub 2020 Mar 4. No abstract available. PMID 32145363
- [Background] Stokkermans TJ, Falkowitz DM, Trichonas G. Chloroquine and Hydroxychloroquine Toxicity. 2024 Jan 11. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK537086/ PMID 30725771
- [Background] Baden LR, Rubin EJ. Covid-19 - The Search for Effective Therapy. N Engl J Med. 2020 May 7;382(19):1851-1852. doi: 10.1056/NEJMe2005477. Epub 2020 Mar 18. No abstract available. PMID 32187463
- [Background] Zhou D, Dai SM, Tong Q. COVID-19: a recommendation to examine the effect of hydroxychloroquine in preventing infection and progression. J Antimicrob Chemother. 2020 Jul 1;75(7):1667-1670. doi: 10.1093/jac/dkaa114. PMID 32196083
- [Background] Chan KW, Wong VT, Tang SCW. COVID-19: An Update on the Epidemiological, Clinical, Preventive and Therapeutic Evidence and Guidelines of Integrative Chinese-Western Medicine for the Management of 2019 Novel Coronavirus Disease. Am J Chin Med. 2020;48(3):737-762. doi: 10.1142/S0192415X20500378. Epub 2020 Mar 13. PMID 32164424
- [Background] Dong L, Hu S, Gao J. Discovering drugs to treat coronavirus disease 2019 (COVID-19). Drug Discov Ther. 2020;14(1):58-60. doi: 10.5582/ddt.2020.01012. PMID 32147628
- [Background] Beigelman A, Bacharier LB, Baty J, Buller R, Mason S, Schechtman KB, Sajol G, Isaacson-Schmid M, Castro M, Storch GA. Does azithromycin modify viral load during severe respiratory syncytial virus bronchiolitis? J Allergy Clin Immunol. 2015 Oct;136(4):1129-31. doi: 10.1016/j.jaci.2015.06.011. Epub 2015 Jul 26. No abstract available. PMID 26215052
- [Background] Jiang S. Don't rush to deploy COVID-19 vaccines and drugs without sufficient safety guarantees. Nature. 2020 Mar;579(7799):321. doi: 10.1038/d41586-020-00751-9. No abstract available. PMID 32179860
- [Background] Cascella M, Rajnik M, Aleem A, Dulebohn SC, Di Napoli R. Features, Evaluation, and Treatment of Coronavirus (COVID-19). 2023 Aug 18. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK554776/ PMID 32150360
- [Background] Fedson DS, Opal SM, Rordam OM. Hiding in Plain Sight: an Approach to Treating Patients with Severe COVID-19 Infection. mBio. 2020 Mar 20;11(2):e00398-20. doi: 10.1128/mBio.00398-20. PMID 32198163
- [Background] Petri M, Elkhalifa M, Li J, Magder LS, Goldman DW. Hydroxychloroquine Blood Levels Predict Hydroxychloroquine Retinopathy. Arthritis Rheumatol. 2020 Mar;72(3):448-453. doi: 10.1002/art.41121. Epub 2020 Jan 7. PMID 31532077
- [Background] Sun ML, Yang JM, Sun YP, Su GH. [Inhibitors of RAS Might Be a Good Choice for the Therapy of COVID-19 Pneumonia]. Zhonghua Jie He He Hu Xi Za Zhi. 2020 Mar 12;43(3):219-222. doi: 10.3760/cma.j.issn.1001-0939.2020.03.016. Chinese. PMID 32164092
- [Background] Sun Q, Qiu H, Huang M, Yang Y. Lower mortality of COVID-19 by early recognition and intervention: experience from Jiangsu Province. Ann Intensive Care. 2020 Mar 18;10(1):33. doi: 10.1186/s13613-020-00650-2. No abstract available. PMID 32189136
- [Background] FitzGerald GA. Misguided drug advice for COVID-19. Science. 2020 Mar 27;367(6485):1434. doi: 10.1126/science.abb8034. Epub 2020 Mar 20. No abstract available. PMID 32198292
- [Background] Lotery A, Burdon M. Monitoring for hydroxychloroquine retinopathy. Eye (Lond). 2020 Aug;34(8):1301-1302. doi: 10.1038/s41433-020-0795-2. Epub 2020 Feb 13. No abstract available. PMID 32055019
- [Background] Devaux CA, Rolain JM, Colson P, Raoult D. New insights on the antiviral effects of chloroquine against coronavirus: what to expect for COVID-19? Int J Antimicrob Agents. 2020 May;55(5):105938. doi: 10.1016/j.ijantimicag.2020.105938. Epub 2020 Mar 12. PMID 32171740
- [Background] Sivakumar GK, Liu J, Sokoluk C, Ing EB. Online calculator for hydroxychloroquine dosing. Can J Ophthalmol. 2020 Aug;55(4):e148-e150. doi: 10.1016/j.jcjo.2020.01.002. Epub 2020 Feb 18. No abstract available. PMID 32081373
- [Background] Guo YR, Cao QD, Hong ZS, Tan YY, Chen SD, Jin HJ, Tan KS, Wang DY, Yan Y. The origin, transmission and clinical therapies on coronavirus disease 2019 (COVID-19) outbreak - an update on the status. Mil Med Res. 2020 Mar 13;7(1):11. doi: 10.1186/s40779-020-00240-0. PMID 32169119
- [Background] Liu F, Xu A, Zhang Y, Xuan W, Yan T, Pan K, Yu W, Zhang J. Patients of COVID-19 may benefit from sustained Lopinavir-combined regimen and the increase of Eosinophil may predict the outcome of COVID-19 progression. Int J Infect Dis. 2020 Jun;95:183-191. doi: 10.1016/j.ijid.2020.03.013. Epub 2020 Mar 12. PMID 32173576
- [Background] Glauser W. Proposed protocol to keep COVID-19 out of hospitals. CMAJ. 2020 Mar 9;192(10):E264-E265. doi: 10.1503/cmaj.1095852. No abstract available. PMID 32152059
- [Background] Baron SA, Devaux C, Colson P, Raoult D, Rolain JM. Teicoplanin: an alternative drug for the treatment of COVID-19? Int J Antimicrob Agents. 2020 Apr;55(4):105944. doi: 10.1016/j.ijantimicag.2020.105944. Epub 2020 Mar 13. PMID 32179150
- [Background] Cunningham AC, Goh HP, Koh D. Treatment of COVID-19: old tricks for new challenges. Crit Care. 2020 Mar 16;24(1):91. doi: 10.1186/s13054-020-2818-6. No abstract available. PMID 32178711
- [Background] Cao B, Wang Y, Wen D, Liu W, Wang J, Fan G, Ruan L, Song B, Cai Y, Wei M, Li X, Xia J, Chen N, Xiang J, Yu T, Bai T, Xie X, Zhang L, Li C, Yuan Y, Chen H, Li H, Huang H, Tu S, Gong F, Liu Y, Wei Y, Dong C, Zhou F, Gu X, Xu J, Liu Z, Zhang Y, Li H, Shang L, Wang K, Li K, Zhou X, Dong X, Qu Z, Lu S, Hu X, Ruan S, Luo S, Wu J, Peng L, Cheng F, Pan L, Zou J, Jia C, Wang J, Liu X, Wang S, Wu X, Ge Q, He J, Zhan H, Qiu F, Guo L, Huang C, Jaki T, Hayden FG, Horby PW, Zhang D, Wang C. A Trial of Lopinavir-Ritonavir in Adults Hospitalized with Severe Covid-19. N Engl J Med. 2020 May 7;382(19):1787-1799. doi: 10.1056/NEJMoa2001282. Epub 2020 Mar 18. PMID 32187464

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Subjects in this arm will receive the study drug
  Hydroxychloroquine: Hydroxychloroquine 800 mg initial dose then 6-8 hours later HCQ 600 mg, then 200 mg three times per day for 4 days.
- Control: Subjects in this arm will take placebo for 6 days
  Placebo: Placebo take 4 tabs, then 6-8 hours later take 3 tabs, then take 1 tab three times per day for 4 days.
Period: Overall Study
Arm/Group | Treatment | Control
Started | 1 | 2
Completed | 1 | 1
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Are Virus Free
Description: Nasopharyngeal swab PCR measurement of viral load expressed as the % of negative PCR swabs
Time Frame: 7 days after initiation of trial
Measure: Number; unit: participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 1 | 1
participants | 0 | 0

2. Primary Outcome: Disease Severity
Description: Participants will self-report disease severity status as one of the following 5 options; no COVID19 illness (score of 1), COVID19 illness with no hospitalization (score of 2), or COVID19 illness with hospitalization (score of 3), or Covid 19 with care requiring hospitalization (score of 4), or Covid 19 with death (Score of 5) .
Time Frame: 6 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 1 | 1
Participants
  no COVID19 illness (score of 1) | 1 | 0
  COVID19 illness with no hospitalization (score of 2) | 0 | 1
  COVID19 illness with hospitalization (score of 3) | 0 | 0
  Covid 19 with care requiring hospitalization (score of 4) | 0 | 0
  Covid 19 with death (Score of 5) | 0 | 0

3. Secondary Outcome: Number of Participants Who Are Hospitalized for Covid 19 Infection
Description: Number of subjects in each arm who are hospitalized for Covid 19 infection
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

4. Secondary Outcome: Number of Participants Who Die Secondary to Covid 19 Infection
Description: Number of subjects in each arm who die secondary to Covid-19 infection
Time Frame: 70 Days (10 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

5. Secondary Outcome: Number of Participants Who Have Confirmed Covid 19 Infection
Description: Number of subjects in each arm who have confirmed Covid-19 infection
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 1 | 2
Participants | 1 | 2

6. Secondary Outcome: Number of Participants Who Discontinue or Withdraw Medication Use for Any Reason
Description: Number of subjects in each arm who discontinue or withdraw medication use for any reason
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 1 | 2
Participants | 0 | 1

7. Secondary Outcome: Immunity to Covid-19
Description: Blood tests to determine level of immunity in each subject
Time Frame: 70 days (10 weeks)
Population: Participants refused blood draw. Data was not collected
Arm/Group | Treatment | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected up to 10 weeks after treatment
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-17): https://cdn.clinicaltrials.gov/large-docs/71/NCT04353271/Prot_SAP_000.pdf